CLINICAL TRIAL: NCT03125876
Title: A Phase Ib, Multi-center, Open, Dose-escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of Ningetinib (CT053PTSA) in Relapsed / Refractory Acute Myeloid Leukemia (AML)
Brief Title: A Phase Ib Study of CT053PTSA in Relapsed / Refractory Acute Myeloid Leukemia (AML)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company strategy adjustment
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCD-DCT053-16-002
Record Dates: First submitted 2017-04-09; First posted 2017-04-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CT053PTSA (Experimental): 60mg-100mg
  Interventions: Drug: CT053PTSA

INTERVENTIONS:
Drug: CT053PTSA — receive oral CT053PTSA once daily until disease progression or unacceptable toxicity occurs, each cycle is defined as 28 days
  Other Names: Ningetinib

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of CT053PTSA in Relapsed/refractory AML patients with FLT3 gene mutation.

DETAILED DESCRIPTION:
It is a multi-center , open-label, dose escalation study conducted in 2 parts. Dose-escalation part: Subjects will receive oral CT053PTSA once daily repeatedly until disease progression or unacceptable toxicity occurs, each cycle is defined as 28 days. At least 3 subjects will receive CT053PTSA at each dose (60, 80, 100mg) for determination of Maximum Tolerated Dose(MTD) and Dose Limiting Toxicity (DLT) Dose reduction of CT053PTSA will be considered if study drug-related toxicities are observed in a subject after Cycle 1.

Expansion part:Expansion cohort might be set to further investigate the safety and efficacy of CT053PTSA at or lower MTD dose recommended by dose-escalation part.

ELIGIBILITY:
Inclusion Criteria:

1. study population

   a) documented acute myeloid leukemia according to World Health Organization（WHO） criteria(excluding acute promyelocytic leukemia), with Fms-like Tyrosine Kinase 3 (FLT3) gene mutation,refractory/relapsed after common or enhanced chemotherapy c) Recovered from toxicity of previous treatment d) Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 e) Life expectation ≥ 12 weeks
2. Subjects must have adequate organ function and meeting all of the following laboratory review before enrollment a)blood routine examination: WBC≤2000/mm3 b)liver function: Alanine aminotransferase (ALT) and Aspartate transaminase (AST) ≤2.5×upper limit of normal(ULN); serum bilirubin ≤ 1.5 × ULN c)renal function: Serum creatinine ≤ 1.5×ULN, or the creatinine clearance (CrCl)≥ 60 mL / min calculated by the Cockcroft-Gault formula d) electrolyte: serum potassium≥3.0mmol/L; serum calcium≥2.0 mmol/L e) abnormal serum amylase without symptom≤1.5 × ULN; serum Lipase ≤1.5× ULN f) coagulation function:fibrinogen≥1.0g/L; activated partial thromboplastin time( APTT)≦ULN+10s; prothrombin time(PT)≤ULN+3s g) no obvious organ dysfunction 3)subjects must volunteer to provide evidence of effective diagnosis prior to entry or to accept bone marrow puncture or biopsy for diagnosis, and accept bone marrow puncture or biopsy after treatment to evaluate the efficacy 4) Sign the informed consent

Exclusion Criteria:

Subject meeting any of the following criteria will be excluded.

1. treatment history

   1. chemotherapy, immunotherapy, radiotherapy, or major surgery within 4 weeks prior to administration;
   2. nitrosourea and mitomycin chemotherapy within 6 weeks prior to the administration;
   3. have taken live vaccines within 4 weeks prior to /or concurrent with the administration;
   4. received FLT3 or Axl inhibitors within 6 weeks prior to the administration;
   5. have received a trial investigational product, or participated in other clinical trials within 4 weeks prior to administration
2. disease history and surgery history

   a) documented promyelocytic leukemia (t (15; 17) (q22; q11) and / or promyelocytic leukemia(PML)/retinoic acid receptor alpha (RARa) positivity found in the chromosome, variant acute promyelocytic leukemia) b) with myeloid sarcoma or invasion of central nervous system; c) high blood pressure and not well controlled by drug (blood pressure ≥ 140/90 mmHg). Note: Blood pressure before the first administration (mean blood pressure of two measures that 24 hours interval or above ) should be controlled within 140/90 mmHg.

   d) Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) <50%; e) NCI CTCAE 4.03 ≥ 2 grade of arrhythmia, or corrected QT interval(QTc )> 450 ms ; patients with a history of torsion or congenital QT prolonged syndrome; f) any of the illness bellowed within 12 months prior to administration: myocardial infarction, severe or unstable angina, coronary artery bypass graft or peripheral artery bypass surgery, congestive heart failure, cerebrovascular events (including Transient ischemic attack); g) multiple factors that affect oral medication (eg, can not swallow, chronic diarrhea and intestinal obstruction, etc.); h)obvious tendency of gastrointestinal bleeding, including the following cases: local active ulcer lesion, and fecal occult blood test(≥++); melena or hematemesis within 2 months; gastrointestinal bleeding may occurs considered by investigator.

   i)history of immunodeficiency, other acquired or congenital immunodeficiency,history of organ transplantation; j) previous thyroid dysfunction,thyroid function can not be maintained at the normal range even have drug taken.

   k)Human immunodeficiency virus(HIV) positivity l) Hepatitis B surface antigen (HBsAg)positivity, and in the active phase(hepatitis B nucleic acid quantity≥ 1.00 × 103copies / ml); m) Hepatitis C antibody(Anti-HCV) positivity and in the active phase (hepatitis C nucleic acid quantity ≥1.00 × 102copies / ml) n) severe retinopathy or exfoliation judged by the Investigator; o) severe electrolyte imbalance judged by the investigator; p) active infectious disease judged by the investigator; q) other acute or chronic medical or psychological illnesses that are not suitable for clinical trials considered by the investigator or sponsor;
3. Pregnant or lactating women or female and male with fertility plan. 4)the therapy and/or drug forbidden

   1. taking anticoagulant or vitamin K antagonist such as warfarin, heparin or other similar drugs;
   2. taking other anti-leukemia drugs at the same time, including traditional Chinese medicine (some Chinese medicine can not be used listed in Annex 4);
   3. taking drugs that will prolong QT interval(including Ia and III antiarrhythmic drugs);
   4. patients who need oxygen therapy every day;
   5. long-term use of corticosteroids (local inhalation excluded);

5)others

a) history of Psychotropic drugs abuse and can not drop or the mentally disordered; b) be used to drink grapefruit juice or too much tea, coffee and / or caffeine-containing drink, can not stop during the trial(including Cycle 1 and subsequent treatment period) c) in the vegistrator's judgment, there is a serious accompany disease that jeopardizes patient's safety or interfere with the completion of the study.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2019-08-19 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | day 1-28
  Safety and Tolerability assessed through adverse events to determine maximum tolerated dose

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | On day 1,8,15,22,29
  to assess the pharmacokinetic profile in patients with AML
Time of maximum observed plasma concentration (Tmax) | On day 1,8,15,22,29
  to assess the pharmacokinetic profile in patients with AML
Area under the plasma concentration time curve | On day 1,8,15,22,29
  to assess the pharmacokinetic profile in patients with AML
Objective response rate (ORR) | Through study completion, an expected average of 1.5 year
  based on investigator review of radiographic images

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, Doctor, Study Chair — Hospital of Blood Disease, Chinese Academy of Medical Sciences
Locations (1):
- Hospital of Blood Disease, Chinese Academy of Medical Sciences, Tianjin, China

IPD SHARING:
Plan to Share IPD: No